CLINICAL TRIAL: NCT00436332
Title: A Phase II Trial of the Combination of OSI-774 (ERLOTINIB; NSC-718781) and Bevacizumab (Rhumab VEGF; NSC-704865) in Stage IIIB and IV Bronchioloalveolar Carcinoma (BAC) and Adenocarcinoma With BAC Features (ADENOBAC)
Brief Title: S0635: Erlotinib and Bevacizumab in Stage IIIB and IV Bronchioloalveolar Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000529756; S0635 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; bronchoalveolar cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib and Bevacizumab (Experimental)
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: bevacizumab
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving erlotinib together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving erlotinib together with bevacizumab works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine overall survival of patients with stage IIIB or IV bronchioloalveolar carcinoma (BAC) or adenocarcinoma with BAC features treated with erlotinib hydrochloride and bevacizumab.

Secondary

* Determine the progression-free survival of patients treated with this regimen.
* Compare, preliminarily, response as assessed by RECIST criteria vs response as assessed by a central computer-assisted image-analysis system in patients with measurable disease treated with this regimen.
* Assess the frequency and severity of toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 2 years.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven* bronchioloalveolar carcinoma (BAC) or BAC variants (e.g., adenocarcinoma with BAC features, BAC with invasive adenocarcinoma) meeting the following criteria:

  * Incompletely resected or unresectable disease
  * No component of squamous cell carcinoma
  * Disease staged as 1 of the following:

    * Stage IIIB disease (T4 [cytologically confirmed malignant pleural effusion OR pleural tumor foci that are separate from direct pleural invasion by the primary tumor], any N, M0)
    * Stage IV disease (any T, any N, M1 [distant metastases present])

      * Recurrent disease in a separate lobe after prior resection within the past 5 years; multifocal lesions in > 1 lobe; or any disease that is recurrent after surgery or radiotherapy is considered stage IV disease
  * Tumor may be multifocal or diffuse NOTE: *Cytology specimens, including bronchial brushing, washings, or fine needle aspiration specimens, alone are not acceptable for diagnosis
* Measurable or nonmeasurable disease by chest CT scan

  * Pleural effusions, ascites, and laboratory parameters are not acceptable as only evidence of disease
  * Disease must be present outside field of prior radiotherapy OR a new lesion must be inside port
* Treated brain metastases allowed provided the patient is asymptomatic and do not require steroids

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal
* AST or AST ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if bone metastases are present)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* Urine protein:creatinine ratio ≤ 0.5 OR urine protein < 1 g by 24-hour urine collection
* Willing to provide prior smoking history
* No hemoptysis ≥ ½ teaspoon within the past 28 days
* No clinical history of pulmonary or upper respiratory hemorrhage > grade 2 within the past 6 months or > grade 1 within the past 28 days
* No history of thromboses or hemorrhage, including hemorrhagic or thrombotic stroke, or other CNS bleeding
* No uncontrolled hypertension
* No serious nonhealing wound, ulcer, or bone fracture
* No other prior malignancy except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer that is currently in complete remission
  * Any other cancer from which the patient has been disease free for 5 years
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 28 days since prior radiotherapy (14 days for palliative radiotherapy)
* At least 28 days since prior surgery (thoracic or other major surgeries)
* More than 7 days since prior fine-needle aspiration or core biopsy
* At least 28 days since prior systemic chemotherapy or biologic therapy
* No prior gefitinib hydrochloride, erlotinib hydrochloride, or bevacizumab
* No other prior anti-epidermal growth factor receptor or anti-vascular endothelial growth factor therapies
* Concurrent stable, therapeutic anticoagulation therapy allowed (i.e., warfarin or low molecular weight heparin), provided the patient has no history of bleeding complications on anticoagulation or an inability to establish a stable therapeutic regimen for anticoagulation
* No other concurrent anticancer therapy, including surgery, chemotherapy, hormone therapy, biologic therapy, or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-07; Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. West, MD, Study Chair — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus
Locations (148):
- United States (148):
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center - Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] West HJ, Moon J, Hirsch FR, et al.: SWOG S0635 and S0636: Phase II trials in advanced-stage NSCLC of erlotinib (OSI-774) and bevacizumab in bronchioloalveolar carcinoma (BAC) and adenocarcinoma with BAC features (adenoBAC), and in never-smokers with primary NSCLC adenocarcinoma (adenoCa). [Abstract] J Clin Oncol 30 (Suppl 15): A-7517, 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib and Bevacizumab: Patients receive 150 mg of erlotinib daily and 15 mg/kg of bevacizumab on day one of the 21-day cycle.
Period: Overall Study
Arm/Group | Erlotinib and Bevacizumab
Started | 84
Eligible | 82
Eligible and Began Protocol Therapy | 79
Completed | 1
Not Completed | 83
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 2
Not completed — Progression | 59
Not completed — Death | 2
Not completed — Not Protocol Specified | 6
Not completed — Ineligible | 2
Not completed — Never Received Treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 79
Age, Continuous [Median (Full Range); unit: years] | 69.2 [39.1 to 92.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 72
  More than one race | 0
  Unknown or Not Reported | 1
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma with Bronchioloalveolar Carcinoma | 56
  Bronchioloalveolar Carcinoma | 23
Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 37
    1 | 39
    2 | 3
Smoking History [Count of Participants; unit: Participants]
  Current | 11
  Former | 61
  Never | 7
Stage [Count of Participants; unit: Participants] — Patients must have selected Stage IIIB disease or Stage IV disease as outlined below (AJCC Cancer Staging Manual, 6th Edition, 2002):
  IIIB
  * T4 (cytology confirmed malignant pleural effusion, OR pleural tumor foci that are separate from direct pleural invasion by the primary tumor)
  * Any N
  * M0
  Stage IV
  * Any T
  * Any N
  * M1 (distant metastases present)
  NOTE: Any disease that is recurrent after surgery or radiation is classified as Stage IV.
  Participants
    IIIB | 3
    IV | 76
Weight Loss Last 6 Months [Count of Participants; unit: Participants]
  <5% | 57
  5-<10% | 8
  10-20% | 10
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: From date of registration to maximum of 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 79
months | 21 [14 to 26]

2. Secondary Outcome: Progression-free Survival
Time Frame: From date of registration to maximum of 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 79
months | 5 [4 to 7]

3. Secondary Outcome: Response as Assessed by RECIST Criteria vs Central Computer-assisted Image-analysis System in Patients With Measurable Disease
Description: Images for response assessed by the central computer-assisted image-analysis system were never collected.
Time Frame: From date of registration to maximum of 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 79
Participants
  Confirmed Complete Response | 2
  Confirmed Partial Response | 5
  Unconfirmed Partial Response | 8
  Stable/No Response | 33
  Progression | 11
  Symptomatic Deterioration | 1
  Early Death | 1
  Assessment Inadequate | 2
  Non Measurable Baseline Disease Status | 16

4. Secondary Outcome: Frequency and Severity of Toxicities
Time Frame: From date of registration to maximum of 3 years
Population: Number of Subjects With Greater Than Grade 2 Toxicity
Measure: Number; unit: participants
Arm/Group | Erlotinib and Bevacizumab
Number analyzed (Participants) | 79
participants
  AST, SGOT | 1
  Albumin, serum-low (hypoalbuminemia) | 1
  Anorexia | 2
  Ataxia (incoordination) | 1
  CNS cerebrovascular ischemia | 3
  Carbon monoxide diffusion capacity (DL(co)) | 1
  Creatinine | 1
  Dehydration | 3
  Diarrhea | 12
  Dry skin | 1
  Dyspnea (shortness of breath) | 2
  Extremity-lower (gait/walking) | 1
  Fatigue (asthenia, lethargy, malaise) | 9
  Hypertension | 6
  Hypoxia | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 2
  Left ventricular diastolic dysfunction | 1
  Left ventricular systolic dysfunction | 1
  Mucositis/stomatitis (clinical exam) - Oral cavity | 1
  Mucositis/stomatitis (functional/symp) - Oral cav | 1
  Muscle weakness, not d/t neuropathy - body/general | 2
  Nail changes | 1
  Nausea | 2
  Ocular/Visual-Other (Specify) | 1
  Pain - Chest wall | 1
  Pain - Extremity-limb | 1
  Pain - Head/headache | 2
  Potassium, serum-high (hyperkalemia) | 1
  Potassium, serum-low (hypokalemia) | 3
  Proteinuria | 3
  Pruritus/itching | 2
  Pulmonary/Upper Respiratory-Other (Specify) | 1
  Rash/desquamation | 5
  Rash: acne/acneiform | 9
  Rash: hand-foot skin reaction | 4
  Renal failure | 1
  Renal/Genitourinary-Other (Specify) | 1
  Retinal detachment | 1
  Sodium, serum-low (hyponatremia) | 2
  Speech impairment (e.g., dysphasia or aphasia) | 1
  Syncope (fainting) | 1
  Ulcer, GI - Duodenum | 1
  Ulcer, GI - Stomach | 1
  Ulceration | 1
  Vomiting | 1
  Weight loss | 3
  Wound complication, non-infectious | 1

ADVERSE EVENTS:
Time Frame: From date of registration to maximum of 3 years.
Description: Only adverse events and serious adverse events that are possibly, probably or definitely related to study drug are reported.
Groups:
- Erlotinib and Bevacizumab: Patients receive oral erlotinib hydrochloride once daily on days 1-21 and bevacizumab IV over 30-90 minutes on day 1.
Arm/Group | Erlotinib and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 56/79
Serious Adverse Events (participants affected / at risk) | 6/79
Other Adverse Events (participants affected / at risk) | 77/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Bevacizumab (N=79)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Retinal detachment (Eye disorders) | 1
Ulcer, GI - Stomach (Gastrointestinal disorders) | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1
Creatinine (Investigations) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Bevacizumab (N=79)
Hemoglobin (Blood and lymphatic system disorders) | 15
Dry eye syndrome (Eye disorders) | 6
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 56
Heartburn/dyspepsia (Gastrointestinal disorders) | 11
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 13
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 31
Vomiting (Gastrointestinal disorders) | 12
Edema: limb (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 55
Rigors/chills (General disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 11
AST, SGOT (Investigations) | 18
Alkaline phosphatase (Investigations) | 8
Bilirubin (hyperbilirubinemia) (Investigations) | 18
Creatinine (Investigations) | 14
Leukocytes (total WBC) (Investigations) | 4
Metabolic/Laboratory-Other (Investigations) | 6
Weight loss (Investigations) | 29
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 28
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 8
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 13
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 7
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 8
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 7
Neuropathy: sensory (Nervous system disorders) | 7
Pain - Head/headache (Nervous system disorders) | 9
Taste alteration (dysgeusia) (Nervous system disorders) | 15
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 17
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 26
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 18
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 23
Nail changes (Skin and subcutaneous tissue disorders) | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 18
Rash/desquamation (Skin and subcutaneous tissue disorders) | 28
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 58
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 11
Hypertension (Vascular disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-12-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT00436332/Prot_SAP_ICF_000.pdf